CLINICAL TRIAL: NCT06676956
Title: The SEQUENCE Trial: Should Endobronchial Ultrasound QUeue bEfore or eNsuing to robotiC-assisted Bronchoscopy for pEripheral Pulmonary Nodule Biopsy? A Patient Randomized Control Trial Assessing the Effect of the Ordering of Robotic-assisted Bronchoscopy and Linear EBUS During the Same Anesthesia Event on Diagnostic Yield From Peripheral Pulmonary Nodule Biopsy
Brief Title: The SEQUENCE Trial: Evaluating Diagnostic Yield of Robotic-assisted Bronchoscopy When Staging EBUS is Performed First or Second in the Same Procedure
Acronym: SEQUENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christopher Kapp, Assistant Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00222248 (IRB)
Record Dates: First submitted 2024-10-28; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Linear EBUS First (Active Comparator): Patients will undergo a mediastinal lymph node evaluation with EBUS first, followed by biopsy followed by robotic-assisted bronchoscopy
  Interventions: Procedure: Order of bronchoscopy procedures for peripheral nodule biopsy
- Robotic-assisted bronchoscopy first (Active Comparator): Patients will undergo a robotic-assisted bronchoscopy first, followed by a mediastinal lymph node evaluation with EBUS second
  Interventions: Procedure: Order of bronchoscopy procedures for peripheral nodule biopsy

INTERVENTIONS:
Procedure: Order of bronchoscopy procedures for peripheral nodule biopsy — Patient scheduled to undergo peripheral nodule biopsy of the lung under bronchoscopy typically get both a nodule biopsy as well as a linear EBUS of the lymph nodes to assess for any disease spread. This procedure will randomize patients to either getting the peripheral nodule first or linear EBUS of the lymph nodes first and assess overall diagnostic yield as the primary outcome.

SUMMARY:
Robotic-assisted bronchoscopy (RaB) has afforded proceduralists the ability to accurately reach the periphery of the lung for biopsy of pulmonary nodules1. This has paved the way for patients to undergo both biopsy of a peripheral nodule and a staging linear endobronchial ultrasound (EBUS) in the same anesthesia event, promoting quicker throughput from discovery of a lesion to guideline-adherent treatment2. Further, introduction and mainstream utilization of cone-beam CT (CBCT) has provided the bronchoscopist the ability to refine needle position with tool-in-lesion confirmation3. While there are no randomized clinical trials promoting efficacy of RaB and CBCT in comparison with other bronchoscopic methods, in single center retrospective studies, diagnostic yield has consistently proven to be in the 70-85% range, superior to prior technologies4-6.

One of the limitations of utilization of RaB and CBCT is the detrimental effect that atelectasis plays in the bronchoscopy procedure. This can lead to false positive radial EBUS (rEBUS) signals and non-diagnostic procedures7. This incidence of atelectasis has been evaluated prospectively, using a protocol featuring 8-10 cmH2O of PEEP and limiting hyperoxia8, and results suggest this ventilator strategy does an adequate job preventing intraprocedural lung collapse. However, this study only evaluated incidence of atelectasis and did not elaborate on its impact on diagnostic yield.

Further unknown is the optimal sequence of performance of RaB and a staging linear EBUS in patients with a radiographically normal mediastinum. Starting with either the RaB or Linear EBUS both have their pros and cons. The benefit to performance of a linear EBUS first is the potential to obviate the need for peripheral nodule biopsy by obtaining rapid, on-site pathologic feedback of occult nodal disease, reducing some of the risk of the procedure (i.e. bleeding and pneumothorax).6 Conversely, the pitfalls to performing linear EBUS first is the possible contribution of atelectasis resultant of the increased time from intubation to peripheral nodule biopsy, blood in the airway causing bronchospasm, and resorption atelectasis from hyperoxia9. There are no prospective data evaluating this in a randomized fashion, but one Monte Carlo simulation (with assumption of diagnostic yield from navigational bronchoscopy of 70% when performed first and 60% when performed second) suggested a higher diagnostic yield and less need for repeat procedure in the navigation first group, despite a 10% assumption of occult nodal disease10.

As outlined in the specific aims above, the overarching goals of this study are to assess in a multicenter, randomized clinical trial performed by members of the Interventional Pulmonary Outcomes Group (IPOG), whether sequence of staging EBUS plays a role in diagnostic yield, incidence of atelectasis, and safety outcomes in patients undergoing RaB.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Pulmonary Nodule undergoing a robotic-assisted bronchoscopy

Exclusion Criteria:

* lymph nodes that are enlarged or PET avid on CT prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield from the procedure | This will be assessed 30 days after the procedure in a study visit that our teams conduct, it will not include the patient
  This will be an outcome measure that is positive or negative based on whether a diagnosis was achieved during the procedure

SECONDARY OUTCOMES:
Atelectasis | This will be assessed day of procedure and recorded
  Using the IPOG atelectasis score (three outcomes) we will track the impact atelectasis has on the biopsy and diagnostic yield

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and collected in a secure REDCap database where only the lead site has access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10/28/24 - two years
Access Criteria: Only study personnel.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT06676956/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT06676956/ICF_001.pdf